CLINICAL TRIAL: NCT04269239
Title: Effectiveness of Healthy Habits for Hospitalized Older Adults to Optimize Rehabilitation
Acronym: HH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sara Nowakowski, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H - 45617 HealthyHab
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Insomnia; Pain; Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Knee Arthroplasty; Hip Arthroplasty; Rehabilitation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain; Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Sleep

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either the a healthy habits group or a sleep habits group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Habits (Other): This group will meet with a study therapist to discuss strategies to implement healthy habits that may enhance recovery from knee or hip surgery.
  Interventions: Behavioral: Healthy Habits
- Sleep Habits (Other): This group will meet with a study therapist to discuss strategies to implement healthy sleep habits that may enhance recovery from knee or hip surgery.
  Interventions: Behavioral: Sleep Habits

INTERVENTIONS:
Behavioral: Healthy Habits — Participants in this group will be coached during four hour-long sessions on topics such as physical activity, nutrition, pain coping skills, bladder health, diabetes, heart health, eyes/vision, hearing, and doctor-patient communication.
  Arms: Healthy Habits
Behavioral: Sleep Habits — Participants in this group will be coached during four hour-long sessions on topics such as sleep education, sleep restriction, stimulus control, cognitive restructuring, sleep hygiene education, and relapse prevention.
  Arms: Sleep Habits

SUMMARY:
This study aims to evaluate behavioral interventions in conjunction with medical rehabilitation to promote functional health in patients recovering from orthopedic surgery. Half of the subjects in this study will be assigned to an intervention that meets with a study therapist to discuss implementing healthy habits. The other half of subjects will assigned to an intervention group that meets with a study therapists to discuss implementing healthy sleep habits. Both groups will undergo several physical and cognitive assessments.

DETAILED DESCRIPTION:
Improving healthy habits such as sleep, nutrition or physical activity is expected to enhance rehabilitation in knee or hip arthroplasty patients, by increasing their ability to attend and adhere to rehabilitation recommendations following surgery. Half of the subjects in this study will be assigned to an intervention that meets with a study therapist to discuss implementing healthy habits (physical activity, nutrition, pain-coping techniques, etc). The other half of subjects will assigned to an intervention group that meets with a study therapists to discuss implementing healthy sleep habits. Both groups will undergo several physical and cognitive assessments at baseline (prior to surgery), post-hospital, post-intervention and at a 6 month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a minimum age of 40 years, no maximum age limit, planning on having a hip or knee arthroplasty.
2. The ability to communicate during the screening process (e.g., no aphasia or other severe language impairment).
3. Meet DSM-5 criteria for insomnia disorder assessed by Duke Structured Interview for Sleep Disorders.
4. Score ≥8 on the Insomnia Severity Index (ISI) or ≥5 on the Pittsburgh Sleep Quality Index (PSQI).
5. Referral and attendance of medical rehabilitation post-discharge.

Exclusion Criteria:

1. Evidence of recent severe mental health disorders (e.g., suicide attempt or psychiatric hospitalization in the past year).
2. Presence of psychotic disorder, substance abuse or dependence, or bipolar disorder assessed by MINI International Neuropsychiatric Inventory (to increase generalizability other psychiatric comorbidities such as depression or anxiety will not be excluded).
3. Untreated comorbid sleep disorders based on structured diagnostic interview including: narcolepsy, periodic leg movement disorder, and/or obstructive sleep apnea risk.
4. Cognitive impairment defined as <20 on the Mini Mental Status Exam (MMSE) that could potentially limit comprehension of the intervention. Note, while an MMSE of <24 is often used as a cutoff for cognitive impairment, we do not wish to exclude those with mild cognitive problems from this study as there is evidence that individuals with mild cognitive problems still benefit from insomnia treatments.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 7-14 days before scheduled surgery
  ISI is a questionnaire that provides a clinically meaningful index of insomnia. It is a 7-item validated self-report scale that assesses subjective symptoms of insomnia. Items are scored on a 0-4 scale to yield a score of 0-28. Higher scores indicate greater insomnia severity. A cutoff score of ≥ 8 is optimal to detect clinical levels of insomnia.
Insomnia Severity Index (ISI) | 7-14 days after hospital discharge
  ISI is a questionnaire that provides a clinically meaningful index of insomnia. It is a 7-item validated self-report scale that assesses subjective symptoms of insomnia. Items are scored on a 0-4 scale to yield a score of 0-28. Higher scores indicate greater insomnia severity. A cutoff score of ≥ 8 is optimal to detect clinical levels of insomnia.
Insomnia Severity Index (ISI) | 7-14 days after completing the 8 week intervention period
  ISI is a questionnaire that provides a clinically meaningful index of insomnia. It is a 7-item validated self-report scale that assesses subjective symptoms of insomnia. Items are scored on a 0-4 scale to yield a score of 0-28. Higher scores indicate greater insomnia severity. A cutoff score of ≥ 8 is optimal to detect clinical levels of insomnia.
Insomnia Severity Index (ISI) | 6 months after completing the intervention
  ISI is a questionnaire that provides a clinically meaningful index of insomnia. It is a 7-item validated self-report scale that assesses subjective symptoms of insomnia. Items are scored on a 0-4 scale to yield a score of 0-28. Higher scores indicate greater insomnia severity. A cutoff score of ≥ 8 is optimal to detect clinical levels of insomnia.
Wrist actigraphy | 7-14 days before scheduled surgery
  A wearable device will be used to measure participant sleep over seven days.
Wrist actigraphy | 7-14 days after hospital discharge
  A wearable device will be used to measure participant sleep over seven days.
Wrist actigraphy | 7-14 days after completing the 8 week intervention period
  A wearable device will be used to measure participant sleep over seven days.
Wrist actigraphy | 6 months after completing the intervention
  A wearable device will be used to measure participant sleep over seven days.

SECONDARY OUTCOMES:
PROMIS Physical Function (short form) | 7-14 days before scheduled surgery
  The PROMIS physical function short form is a 10 item questionnaire used to assess patient perceived motor abilities. Participants are asked five questions to rank 'from not at all' to 'cannot do' how their health limits their involvement in different activities. Five additional questions ask participants if they are able to complete activities of daily living ranked from 'without any difficulty' to 'unable to do'
PROMIS Physical Function (short form) | 7-14 days after hospital discharge
  The PROMIS physical function short form is a 10 item questionnaire used to assess patient perceived motor abilities. Participants are asked five questions to rank 'from not at all' to 'cannot do' how their health limits their involvement in different activities. Five additional questions ask participants if they are able to complete activities of daily living ranked from 'without any difficulty' to 'unable to do'
PROMIS Physical Function (short form) | 7-14 days after completing the 8 week intervention period
  The PROMIS physical function short form is a 10 item questionnaire used to assess patient perceived motor abilities. Participants are asked five questions to rank 'from not at all' to 'cannot do' how their health limits their involvement in different activities. Five additional questions ask participants if they are able to complete activities of daily living ranked from 'without any difficulty' to 'unable to do'
PROMIS Physical Function (short form) | 6 months after completing the intervention
  The PROMIS physical function short form is a 10 item questionnaire used to assess patient perceived motor abilities. Participants are asked five questions to rank 'from not at all' to 'cannot do' how their health limits their involvement in different activities. Five additional questions ask participants if they are able to complete activities of daily living ranked from 'without any difficulty' to 'unable to do'
PROMIS Mobility | 7-14 days before scheduled surgery
  The PROMIS Mobility questionnaire has 14 questions also used to used to assess patient perceived motor abilities. Participants are asked to respond on a five-point scale from 'without any difficulty' to 'unable to do' about their ability to perform various physical activities.
PROMIS Mobility | 7-14 days after hospital discharge
  The PROMIS Mobility questionnaire has 14 questions also used to used to assess patient perceived motor abilities. Participants are asked to respond on a five-point scale from 'without any difficulty' to 'unable to do' about their ability to perform various physical activities.
PROMIS Mobility | 7-14 days after completing the 8 week intervention period
  The PROMIS Mobility questionnaire has 14 questions also used to used to assess patient perceived motor abilities. Participants are asked to respond on a five-point scale from 'without any difficulty' to 'unable to do' about their ability to perform various physical activities.
PROMIS Mobility | 6 months after completing the intervention
  The PROMIS Mobility questionnaire has 14 questions also used to used to assess patient perceived motor abilities. Participants are asked to respond on a five-point scale from 'without any difficulty' to 'unable to do' about their ability to perform various physical activities.
Short Physical Performance Battery (SPPB ) motor | 7-14 days before scheduled surgery
  The Short Physical Performance Battery (SPPB ) is an objective assessment tool for evaluating lower extremity functioning, developed by the NIA. Motor tests include: a chair stand test, standing balance test (side by side stand, semi-tandem stand, tandem stand.),and gait speed test. The three motor tests are scored and a global score is obtained.
Short Physical Performance Battery (SPPB ) motor | 7-14 days after hospital discharge
  The Short Physical Performance Battery (SPPB ) is an objective assessment tool for evaluating lower extremity functioning, developed by the NIA. Motor tests include: a chair stand test, standing balance test (side by side stand, semi-tandem stand, tandem stand.),and gait speed test. The three motor tests are scored and a global score is obtained.
Short Physical Performance Battery (SPPB ) motor | 7-14 days after completing the 8 week intervention period
  The Short Physical Performance Battery (SPPB ) is an objective assessment tool for evaluating lower extremity functioning, developed by the NIA. Motor tests include: a chair stand test, standing balance test (side by side stand, semi-tandem stand, tandem stand.),and gait speed test. The three motor tests are scored and a global score is obtained.
Short Physical Performance Battery (SPPB ) motor | 6 months after completing the intervention
  The Short Physical Performance Battery (SPPB ) is an objective assessment tool for evaluating lower extremity functioning, developed by the NIA. Motor tests include: a chair stand test, standing balance test (side by side stand, semi-tandem stand, tandem stand.),and gait speed test. The three motor tests are scored and a global score is obtained.
PROMIS Applied Cognitive Abilities | 7-14 days before scheduled surgery
  The PROMIS Applied Cognitive Abilities is a 8 item questionnaire used to assess patient perceived cognitive abilities based on self-report. Participants are asked to rank on a 5 point scale from 'not at all' to 'very much' their perceived cognitive performance over the past seven days.
PROMIS Applied Cognitive Abilities | 7-14 days after hospital discharge
  The PROMIS Applied Cognitive Abilities is a 8 item questionnaire used to assess patient perceived cognitive abilities based on self-report. Participants are asked to rank on a 5 point scale from 'not at all' to 'very much' their perceived cognitive performance over the past seven days.
PROMIS Applied Cognitive Abilities | 7-14 days after completing the 8 week intervention period
  The PROMIS Applied Cognitive Abilities is a 8 item questionnaire used to assess patient perceived cognitive abilities based on self-report. Participants are asked to rank on a 5 point scale from 'not at all' to 'very much' their perceived cognitive performance over the past seven days.
PROMIS Applied Cognitive Abilities | 6 months after completing the intervention
  The PROMIS Applied Cognitive Abilities is a 8 item questionnaire used to assess patient perceived cognitive abilities based on self-report. Participants are asked to rank on a 5 point scale from 'not at all' to 'very much' their perceived cognitive performance over the past seven days.
PROMIS Applied Cognitive Abilities- General Concerns | 7-14 days before scheduled surgery
  The PROMIS Applied Cognitive Abilities is a 6 item questionnaire also used to assess patient perceived cognitive abilities based on self-report. Participants are asked to rank on a five point scale from 'never' to 'very often' the incidence of perceived cognitive impairment over the past seven days.
PROMIS Applied Cognitive Abilities- General Concerns | 7-14 days after hospital discharge
  The PROMIS Applied Cognitive Abilities is a 6 item questionnaire also used to assess patient perceived cognitive abilities based on self-report. Participants are asked to rank on a five point scale from 'never' to 'very often' the incidence of perceived cognitive impairment over the past seven days.
PROMIS Applied Cognitive Abilities- General Concerns | 7-14 days after completing the 8 week intervention period
  The PROMIS Applied Cognitive Abilities is a 6 item questionnaire also used to assess patient perceived cognitive abilities based on self-report. Participants are asked to rank on a five point scale from 'never' to 'very often' the incidence of perceived cognitive impairment over the past seven days.
PROMIS Applied Cognitive Abilities - General Concerns | 6 months after completing the intervention
  The PROMIS Applied Cognitive Abilities is a 6 item questionnaire also used to assess patient perceived cognitive abilities based on self-report. Participants are asked to rank on a five point scale from 'never' to 'very often' the incidence of perceived cognitive impairment over the past seven days.
Tele-neuropsychology (T-NP) Battery | 7-14 days before scheduled surgery
  The T-NP Battery consists of cognitive tests which measure verbal memory, verbal and phonemic fluency, working memory (list sorting, list learning, delayed recall) Cognition tests will be scored.
Tele-neuropsychology (T-NP) Battery | 7-14 days after hospital discharge
  The T-NP Battery consists of cognitive tests which measure verbal memory, verbal and phonemic fluency, working memory (list sorting, list learning, delayed recall). Cognition tests will be scored.
Tele-neuropsychology (T-NP) Battery | 7-14 days after completing the 8 week intervention period
  The T-NP Battery consists of cognitive tests which measure verbal memory, verbal and phonemic fluency, working memory (list sorting, list learning, delayed recall). Cognition tests will be scored.
Tele-neuropsychology (T-NP) Battery | 6 months after completing the intervention
  The TNP Battery consists of cognitive tests which measure verbal memory, verbal and phonemic fluency, working memory (list sorting, list learning, delayed recall). Cognition tests will be scored.
Activities of Daily Living (ADLs) | 7-14 days before scheduled surgery
  The ADL questionnaire measure self-reported activities of daily living (ADLs). The questionnaire assesses need for assistance in 7 activities of daily living (i.e., eating, dressing, grooming, mobility, transferring, bathing, and continence) - questions are answered as "need help" or "don't need help"
Activities of Daily Living (ADLs) | 7-14 days after hospital discharge
  The ADL questionnaire measure self-reported activities of daily living (ADLs). The questionnaire assesses need for assistance in 7 activities of daily living (i.e., eating, dressing, grooming, mobility, transferring, bathing, and continence) - questions are answered as "need help" or "don't need help"
Activities of Daily Living (ADLs) | 7-14 days after completing the 8 week intervention period
  The ADL questionnaire measure self-reported activities of daily living (ADLs). The questionnaire assesses need for assistance in 7 activities of daily living (i.e., eating, dressing, grooming, mobility, transferring, bathing, and continence) - questions are answered as "need help" or "don't need help"
Activities of Daily Living (ADLs) | 6 months after completing the intervention
  The ADL questionnaire measure self-reported activities of daily living (ADLs). The questionnaire assesses need for assistance in 7 activities of daily living (i.e., eating, dressing, grooming, mobility, transferring, bathing, and continence) - questions are answered as "need help" or "don't need help"
Instrumental ADLs (IADL) scale | 7-14 days before scheduled surgery
  The IADL questionnaire is an 8-item scale designed to assesses the need for assistance in telephone use, shopping, food preparation, housekeeping, laundry, transportation, taking medicines and finances. Higher scores indicate greater independence. The questions are answered in a "yes" or "no" format.
Instrumental ADLs (IADL) scale | 7-14 days after hospital discharge
  The IADL questionnaire is an 8-item scale designed to assesses the need for assistance in telephone use, shopping, food preparation, housekeeping, laundry, transportation, taking medicines and finances. Higher scores indicate greater independence. The questions are answered in a "yes" or "no" format.
Instrumental ADLs (IADL) scale | 7-14 days after completing the 8 week intervention period and
  The IADL questionnaire is an 8-item scale designed to assesses the need for assistance in telephone use, shopping, food preparation, housekeeping, laundry, transportation, taking medicines and finances. Higher scores indicate greater independence. The questions are answered in a "yes" or "no" format.
Instrumental ADLs (IADL) scale | 6 months after completing the intervention
  The IADL questionnaire is an 8-item scale designed to assesses the need for assistance in telephone use, shopping, food preparation, housekeeping, laundry, transportation, taking medicines and finances. Higher scores indicate greater independence. The questions are answered in a "yes" or "no" format.
Sleep Diary | 7-14 days before scheduled surgery
  The sleep diary has 9 core items that query: 1) napping, 2) bedtime, 3) time of first attempt to sleep, 4) time to fall asleep, 5) number of awakenings, 6) duration of awakenings, 7) final wake-up time, 8) rise time, 9) a rating of sleep quality, and an optional space for writing comments.
Sleep Diary | 7-14 days after hospital discharge
  The sleep diary has 9 core items that query: 1) napping, 2) bedtime, 3) time of first attempt to sleep, 4) time to fall asleep, 5) number of awakenings, 6) duration of awakenings, 7) final wake-up time, 8) rise time, 9) a rating of sleep quality, and an optional space for writing comments.
Sleep Diary | During the 8 week intervention
  The sleep diary has 9 core items that query: 1) napping, 2) bedtime, 3) time of first attempt to sleep, 4) time to fall asleep, 5) number of awakenings, 6) duration of awakenings, 7) final wake-up time, 8) rise time, 9) a rating of sleep quality, and an optional space for writing comments.
Sleep Diary | 7-14 days after completing the 8 week intervention period
  The sleep diary has 9 core items that query: 1) napping, 2) bedtime, 3) time of first attempt to sleep, 4) time to fall asleep, 5) number of awakenings, 6) duration of awakenings, 7) final wake-up time, 8) rise time, 9) a rating of sleep quality, and an optional space for writing comments.
Sleep Diary | 6 months after completing the intervention
  The sleep diary has 9 core items that query: 1) napping, 2) bedtime, 3) time of first attempt to sleep, 4) time to fall asleep, 5) number of awakenings, 6) duration of awakenings, 7) final wake-up time, 8) rise time, 9) a rating of sleep quality, and an optional space for writing comments.
Knee injury and osteoarthritis outcome score (KOOS) | 7-14 days before scheduled surgery
  This questionnaire is divided into subscales of pain, symptoms, activities of daily living, sports/recreation and quality of life. Questions about how knee pain affects participant in each of these categories answered on a scale of None, Mild, Moderate, Severe or Extremely.
Knee injury and osteoarthritis outcome score (KOOS) | 6 months after completing intervention
  This questionnaire is divided into subscales of pain, symptoms, activities of daily living, sports/recreation and quality of life. Questions about how knee pain affects participant in each of these categories answered on a scale of None, Mild, Moderate, Severe or Extremely.
Hip disability and osteoarthritis outcome score (HOOS) | 7-14 days before scheduled surgery
  This questionnaire is divided into subscales of pain, symptoms, activities of daily living, sports/recreation and quality of life. Questions about how hip pain affects participant in each of these categories answered on a scale of None, Mild, Moderate, Severe or Extremely.
Hip disability and osteoarthritis outcome score (HOOS) | 6 months after completing intervention
  This questionnaire is divided into subscales of pain, symptoms, activities of daily living, sports/recreation and quality of life. Questions about how hip pain affects participant in each of these categories answered on a scale of None, Mild, Moderate, Severe or Extremely.
StepWatch | 7-14 days before scheduled surgery
  A wearable device will measure physical activity over a seven day period.
StepWatch | 7-14 days after hospital discharge
  A wearable device will measure physical activity over a seven day period.
StepWatch | 7-14 days after completing the 8 week intervention period
  A wearable device will measure physical activity over a seven day period.
StepWatch | 6 months after completing the intervention
  A wearable device will measure physical activity over a seven day period.

OTHER OUTCOMES:
PROMIS Pain Intensity | 7-14 days before scheduled surgery
  The PROMIS Pain Intensity is a 3 question questionnaire that asks participants to rank intensity of past and current pain over the last seven days on a five point scale from 'had no pain' to 'very severe'.
PROMIS Pain Intensity | 7-14 days after hospital discharge
  The PROMIS Pain Intensity is a 3 question questionnaire that asks participants to rank intensity of past and current pain over the last seven days on a five point scale from 'had no pain' to 'very severe'.
PROMIS Pain Intensity | 7-14 days after completing the 8 week intervention period
  The PROMIS Pain Intensity is a 3 question questionnaire that asks participants to rank intensity of past and current pain over the last seven days on a five point scale from 'had no pain' to 'very severe'.
PROMIS Pain Intensity | 6 months after completing the intervention
  The PROMIS Pain Intensity is a 3 question questionnaire that asks participants to rank intensity of past and current pain over the last seven days on a five point scale from 'had no pain' to 'very severe'.
PROMIS Pain Interference | 7-14 days before schedule surgery
  The PROMIS Pain Interference is a 6 question questionnaire that ask participants to rank how pain interfered with aspects of their daily life on a five point scale from 'not at all' to 'very much'.
PROMIS Pain Interference | 7-14 days after hospital discharge
  The PROMIS Pain Interference is a 6 question questionnaire that ask participants to rank how pain interfered with aspects of their daily life on a five point scale from 'not at all' to 'very much'.
PROMIS Pain Interference | 7-14 days after completing the 8 week intervention period
  The PROMIS Pain Interference is a 6 question questionnaire that ask participants to rank how pain interfered with aspects of their daily life on a five point scale from 'not at all' to 'very much'.
PROMIS Pain Interference | 6 months after completing the intervention
  The PROMIS Pain Interference is a 6 question questionnaire that ask participants to rank how pain interfered with aspects of their daily life on a five point scale from 'not at all' to 'very much'.
PROMIS Fatigue | 7-14 days before scheduled surgery
  The PROMIS Fatigue questionnaire has 8 questions that ask participants on a five point scale of either 'not at all' to very much' or 'never' to 'always' different statements about fatigue and how it impacted their activities of daily living.
PROMIS Fatigue | 7-14 days after hospital discharge
  The PROMIS Fatigue questionnaire has 8 questions that ask participants on a five point scale of either 'not at all' to very much' or 'never' to 'always' different statements about fatigue and how it impacted their activities of daily living.
PROMIS Fatigue | 7-14 days after completing the 8 week intervention period
  The PROMIS Fatigue questionnaire has 8 questions that ask participants on a five point scale of either 'not at all' to very much' or 'never' to 'always' different statements about fatigue and how it impacted their activities of daily living.
PROMIS Fatigue | 6 months after completing the intervention
  The PROMIS Fatigue questionnaire has 8 questions that ask participants on a five point scale of either 'not at all' to very much' or 'never' to 'always' different statements about fatigue and how it impacted their activities of daily living.
PROMIS Emotional Distress-Depressesion | 7-14 days before scheduled surgery
  The PROMIS Emotional Distress-Depression questionnaire has 8 questions that asks participants to rank on a five point scale form 'never' to 'always' the frequency of different negative feelings over the past seven days.
PROMIS Emotional Distress-Depressesion | 7-14 days after hospital discharge
  The PROMIS Emotional Distress-Depression questionnaire has 8 questions that asks participants to rank on a five point scale form 'never' to 'always' the frequency of different negative feelings over the past seven days.
PROMIS Emotional Distress-Depressesion | 7-14 days after completing the 8 week intervention period
  The PROMIS Emotional Distress-Depression questionnaire has 8 questions that asks participants to rank on a five point scale form 'never' to 'always' the frequency of different negative feelings over the past seven days.
PROMIS Emotional Distress-Depressesion | 6 months after completing the intervention
  The PROMIS Emotional Distress-Depression questionnaire has 8 questions that asks participants to rank on a five point scale form 'never' to 'always' the frequency of different negative feelings over the past seven days.
PROMIS Psychosocial Illness Impact - Negative | 7-14 days before scheduled surgery
  The PROMIS Psychosocial Illness Impact - Negative questionnaire has 16 questions that query participants about 8 aspects of psychosocial well being over the past seven days ranked on a five point scale from 'not at all' to 'very much'.
PROMIS Psychosocial Illness Impact - Negative | 7-14 days after hospital discharge
  The PROMIS Psychosocial Illness Impact - Negative questionnaire has 16 questions that query participants about 8 aspects of psychosocial well being over the past seven days ranked on a five point scale from 'not at all' to 'very much'.
PROMIS Psychosocial Illness Impact - Negative | 7-14 days after completing the 8 week intervention period
  The PROMIS Psychosocial Illness Impact - Negative questionnaire has 16 questions that query participants about 8 aspects of psychosocial well being over the past seven days ranked on a five point scale from 'not at all' to 'very much'.
PROMIS Psychosocial Illness Impact - Negative | 6 months after completing the intervention
  The PROMIS Psychosocial Illness Impact - Negative questionnaire has 16 questions that query participants about 8 aspects of psychosocial well being over the past seven days ranked on a five point scale from 'not at all' to 'very much'.
PROMIS Satisfaction with Social Roles and Activities | 7-14 days before scheduled surgery
  The PROMIS Satisfaction with Social Roles and Activities questionnaire has 4 questions that assess participants satisfaction in their social roles ranked on a five point scale from 'not at all' to 'very much'.
PROMIS Satisfaction with Social Roles and Activities | 7-14 days after hospital discharge
  The PROMIS Satisfaction with Social Roles and Activities questionnaire has 4 questions that assess participants satisfaction in their social roles ranked on a five point scale from 'not at all' to 'very much'.
PROMIS Satisfaction with Social Roles and Activities | 7-14 days after completing the 8 week intervention period
  The PROMIS Satisfaction with Social Roles and Activities questionnaire has 4 questions that assess participants satisfaction in their social roles ranked on a five point scale from 'not at all' to 'very much'.
PROMIS Satisfaction with Social Roles and Activities | 6 months after completing the intervention
  The PROMIS Satisfaction with Social Roles and Activities questionnaire has 4 questions that assess participants satisfaction in their social roles ranked on a five point scale from 'not at all' to 'very much'.
PROMIS Ability to Participate in Social Roles and Activity | 7-14 days before scheduled surgery
  The PROMIS Ability to Participate in Social Roles and Activity questionnaire has four questions that asks participants about their ability to participate socially ranked on a five point scale from 'not at all' to 'very much'.
PROMIS Ability to Participate in Social Roles and Activity | 7-14 days after hospital discharge
  The PROMIS Ability to Participate in Social Roles and Activity questionnaire has four questions that asks participants about their ability to participate socially ranked on a five point scale from 'not at all' to 'very much'.
PROMIS Ability to Participate in Social Roles and Activity | 7-14 days after completing the 8 week intervention period
  The PROMIS Ability to Participate in Social Roles and Activity questionnaire has four questions that asks participants about their ability to participate socially ranked on a five point scale from 'not at all' to 'very much'.
PROMIS Ability to Participate in Social Roles and Activity | 6 months after completing the intervention
  The PROMIS Ability to Participate in Social Roles and Activity questionnaire has four questions that asks participants about their ability to participate socially ranked on a five point scale from 'not at all' to 'very much'.
Rehabilitation Attendance | From hospital discharge until subject notifies study staff they have stopped attending, on average around 12 weeks.
  Weekly rehabilitation attendance will be measured via patient self-report.
Plasma IL-6 | 7-14 days before scheduled surgery
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine Interleukin-6 (IL-6).
Plasma IL-6 | 7-14 days after hospital discharge
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine Interleukin-6 (IL-6).
Plasma IL-6 | 7-14 days after completing the 8 week intervention period
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine Interleukin-6 (IL-6).
Plasma IL-6 | 6 months after completing the intervention
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine Interleukin-6 (IL-6).
Plasma CRP | 7-14 days before scheduled surgery
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine C-reactive protein (CRP)
Plasma CRP | 7-14 days after hospital discharge
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine C-reactive protein (CRP)
Plasma CRP | 7-14 days after completing the 8 week intervention period
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine C-reactive protein (CRP)
Plasma CRP | 6 months after completing the intervention
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine C-reactive protein (CRP)
Plasma VWF | 7-14 days before scheduled surgery
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine vonWillebrand factor (VWF)
Plasma VWF | 7-14 days after hospital discharge
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine vonWillebrand factor (VWF)
Plasma VWF | 7-14 days after completing the 8 week intervention period
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine vonWillebrand factor (VWF)
Plasma VWF | 6 months after completing the intervention
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine vonWillebrand factor (VWF)
Plasma TNFalpha | 7-14 days before scheduled surgery
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine Tumor Necrosis Factor alpha (TNFa)
Plasma TNFalpha | 7-14 days after hospital discharge
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine Tumor Necrosis Factor alpha (TNFa)
Plasma TNFalpha | 7-14 days after completing the 8 week intervention period
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine Tumor Necrosis Factor alpha (TNFa)
Plasma TNFalpha | 6 months after completing the intervention
  Blood samples will be taken by study staff to measure circulating proinflammatory cytokine Tumor Necrosis Factor alpha (TNFa)
Medication Monitoring Form | 7-14 days before schedule surgery
  Medication Monitoring Form will be used to track medication use. Medications will be coded by drug class.
Medication Monitoring Form | 7-14 days after hospital discharge
  Medication Monitoring Form will be used to track medication use. Medications will be coded by drug class.
Medication Monitoring Form | 7-14 days after completing the 8 week intervention period
  Medication Monitoring Form will be used to track medication use. Medications will be coded by drug class.
Medication Monitoring Form | 6 months after completing the intervention
  Medication Monitoring Form will be used to track medication use. Medications will be coded by drug class.
Treatment Expectation Questionnaire | Immediately prior to beginning the intervention
  This questionnaire 8-question measure provided before treatment. It will be used to collect information on participants' reasons for treatment as well as their expectations of treatment (e.g., its effectiveness, the amount of effort it will take, confidence in their doctor). Participant will mark answers to each question on a visual analog scale (e.g., from Not Confident at all to Very Confident).
Treatment Satisfaction Questionnaire | Immediately following the completion of the intervention
  Treatment Satisfaction Scale is a 10-question measure provided after treatment. It measures participants' perceptions on the treatment's effectiveness, benefits, and influence on quality of life (e.g., improvements in work productivity, mood, etc.). Questions are measured on a 5-point Likert scale from Not at all to Very Much.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Nowakowski, PhD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Kelsey Seybold Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: No